CLINICAL TRIAL: NCT02792517
Title: A Multi-Center, Open-label, Pharmacokinetic Drug Interaction Study of AMG 334 and a Combined Oral Contraceptive in Healthy Female Subjects
Brief Title: Erenumab (AMG 334) Plus Combined Oral Contraceptive Drug Interaction Study in Healthy Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20150334
Record Dates: First submitted 2016-02-23; First posted 2016-06-07 (Estimated); Results first posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-05

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erenumab + Estrogen/Progestin Contraceptive (Experimental): Participants received a combination oral contraceptive for 3 28-day cycles during the study.
  A single 140 mg dose of erenumab was administered subcutaneously to the abdomen on day 10 of cycle 3 by a healthcare provider.
  Interventions: Drug: Erenumab; Drug: Ethynil Estradiol/Norgestimate Oral Contraceptive

INTERVENTIONS:
Drug: Erenumab — A single dose of erenumab administered in the abdomen.
  Other Names: AMG-334; Aimovig™
Drug: Ethynil Estradiol/Norgestimate Oral Contraceptive — Ethynil estradiol (EE)/norgestimate combination oral contraceptive is a 28-tablet cycle in which 1 oral tablet is taken daily; each containing 0.250 mg norgestimate and 0.035 mg EE for 21 days, after which a tablet only containing inert ingredients is taken for last 7 days of the 28 day cycle.
  Other Names: Ortho-Cyclen®

SUMMARY:
A pharmacokinetic drug interaction study of erenumab and an oral contraceptive containing progestin and estrogen.

DETAILED DESCRIPTION:
A pharmacokinetic (PK) drug interaction study of erenumab and an oral contraceptive containing progestin and estrogen. All participants will receive an oral contraceptive containing progestin and estrogen throughout the duration of the study. Participants will also receive a single dose of erenumab, administered by a healthcare provider in cycle 3. Serial PK samples will be collected at specified time points to characterize the PK of the oral contraceptive progestin and estrogen components with and without the presence of erenumab.

The study consists of three 28-day cycles and a follow-up period. The first 28 day cycle is an acclimation period when participants initiate oral contraception (Cycle 1). During Cycle 2 and 3 the PK of ethinyl estradiol (EE) and active metabolites of norgestimate (ie, norelgestromin [NGMN] and norgestrel [NG]) will be characterized following the last active dose of oral contraceptive in each cycle (cycle day 21). Erenumab will be given in cycle 3 (cycle day 10); 24-hour PK characterization of norgestimate and EE metabolites will occur 11 days after administration of erenumab, which will maximize the potential for detecting a drug-drug interaction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female ≥18 to ≤45 years old at the time of enrollment
* Regular monthly menstrual cycle during the last 12 months
* Good general health based on a medical history evaluation and physical examination
* No clinically significant abnormalities in laboratory tests at screening
* Subject has provided informed consent/assent prior to initiation of any study specific activities/procedures

Exclusion Criteria:

* Intolerance to any recent oral contraceptive in the last three (3) years,
* Female subjects with a positive serum pregnancy test at screening
* Female subjects not willing to inform her sexual partner of her participation in the clinical study
* Use of any over the counter or prescription medications within the 14 days or 5 half lives (whichever is longer)
* Nicotine use eg cigarettes or equivalent during 12 months prior to day 1 and through the duration of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - Research Site, Anaheim, California
  - Research Site, Cypress, California
  - Research Site, Dallas, Texas
  - Research Site, Madison, Wisconsin

REFERENCES:
- [Derived] Xu Y, Gabriel K, Wang Y, Zhou Y, Eisele O, Vutikullird A, Mikol DD, Lee E. A Multi-Center, Open-Label, Pharmacokinetic Drug Interaction Study of Erenumab and a Combined Oral Contraceptive in Healthy Females. CNS Drugs. 2019 May;33(5):513-522. doi: 10.1007/s40263-019-00626-2. PMID 30963506
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 3 centers in the United States of America. Participants were enrolled from 12 February 2016 to 15 April 2016.
Groups:
- Erenumab 140 mg + Estrogen/Progestin Contraceptive: Participants received a combination oral contraceptive for three 28-day cycles during the study. A single 140 mg dose of erenumab was administered subcutaneously to the abdomen on day 10 of cycle 3 by a healthcare provider.
Period: Overall Study
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Started | 41
Received Erenumab | 24
Completed | 21
Not Completed | 20
Not completed — Withdrawal by Subject | 10
Not completed — Decision by Sponsor | 7
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug (erenumab).
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 10
  Black (or African American) | 6
  Native Hawaiian or Other Pacific Islander | 1
  White | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ethinyl Estradiol
Description: The pharmacokinetics of ethinyl estradiol (EE) were characterized during cycle 2 following the last active dose of oral contraceptive in the cycle (cycle day 21) without erenumab, and during cycle 3 following the last active dose of oral contraceptive in the cycle (cycle day 21), 11 days after a single dose of erenumab.
Time Frame: Cycle 2, day 21 and cycle 3, day 21 at predose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, and 24 hours post oral contraceptive dose.
Population: The pharmacokinetic (PK) analysis set included all participants for whom at least 1 EE, NGMN, and NG PK parameter or endpoint could be adequately estimated. Data are reported for participants with observations at each time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 25
pg/mL
  Cycle 2 (EE/norgestimate alone) | 132 (46.3)
  Cycle 3 (EE/norgestimate with erenumab): number analyzed (Participants) | 22
  Cycle 3 (EE/norgestimate with erenumab) | 143 (64.5)
Statistical Analysis 1: Comparison: Erenumab 140 mg + Estrogen/Progestin Contraceptive; The log-transformed Cmax was analyzed using a linear mixed effects model with treatment as a fixed effect and subject as a random effect; Test type: Other; Least Squares Geometric Mean Ratio = 1.04, 90% CI 2-sided [0.88 to 1.22] — Ratio of EE/norgestimate + erenumab to EE/norgestimate alone

2. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to 24 Hours Postdose (AUCtau) for Ethinyl Estradiol
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL*hr
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 25
pg/mL*hr
  Cycle 2 (EE/norgestimate alone) | 1010 (367)
  Cycle 3 (EE/norgestimate with erenumab): number analyzed (Participants) | 22
  Cycle 3 (EE/norgestimate with erenumab) | 1060 (508)
Statistical Analysis 1: Comparison: Erenumab 140 mg + Estrogen/Progestin Contraceptive; The log-transformed AUCtau was analyzed using a linear mixed effects model with treatment as a fixed effect and subject as a random effect; Test type: Other; Least Squares Geometric Mean Ratio = 1.02, 90% CI 2-sided [0.91 to 1.14] — Ratio of EE/norgestimate + erenumab to EE/norgestimate alone

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Norgestrel
Description: The pharmacokinetics of norgestrel (NG), an active metabolite of norgestimate, were characterized during cycle 2 following the last active dose of oral contraceptive in the cycle (cycle day 21) without erenumab, and during cycle 3 following the last active dose of oral contraceptive in the cycle (cycle day 21), 11 days after a single dose of erenumab.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 25
pg/mL
  Cycle 2 (EE/norgestimate alone) | 2690 (887)
  Cycle 3 (EE/norgestimate with erenumab): number analyzed (Participants) | 22
  Cycle 3 (EE/norgestimate with erenumab) | 2860 (927)
Statistical Analysis 1: Comparison: Erenumab 140 mg + Estrogen/Progestin Contraceptive; [analysis description as in outcome 1, analysis 1]; Test type: Other; Least Squares Geometric Mean Ratio = 1.06, 90% CI 2-sided [0.97 to 1.16] — Ratio of EE/norgestimate + erenumab to EE/norgestimate alone

4. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to 24 Hours Postdose (AUCtau) for Norgestrel
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL*hr
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 25
pg/mL*hr
  Cycle 2 (EE/norgestimate alone) | 50700 (17400)
  Cycle 3 (EE/norgestimate with erenumab): number analyzed (Participants) | 22
  Cycle 3 (EE/norgestimate with erenumab) | 52400 (17400)
Statistical Analysis 1: Comparison: Erenumab 140 mg + Estrogen/Progestin Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Other; Least Squares Geometric Mean Ratio = 1.03, 90% CI 2-sided [0.96 to 1.10] — Ratio of EE/norgestimate + erenumab to EE/norgestimate alone

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Norelgestromin
Description: The pharmacokinetics of norelgestromin (NGMN), an active metabolite of norgestimate, were characterized during cycle 2 following the last active dose of oral contraceptive in the cycle (cycle day 21) without erenumab, and during cycle 3 following the last active dose of oral contraceptive in the cycle (cycle day 21), 11 days after a single dose of erenumab.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 25
pg/mL
  Cycle 2 (EE/norgestimate alone) | 1800 (641)
  Cycle 3 (EE/norgestimate with erenumab): number analyzed (Participants) | 22
  Cycle 3 (EE/norgestimate with erenumab) | 1870 (553)
Statistical Analysis 1: Comparison: Erenumab 140 mg + Estrogen/Progestin Contraceptive; [analysis description as in outcome 1, analysis 1]; Test type: Other; Least Squares Geometric Mean Ratio = 1.05, 90% CI 2-sided [0.90 to 1.23] — Ratio of EE/norgestimate + erenumab to EE/norgestimate alone

6. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to 24 Hours Postdose (AUCtau) for Norelgestromin
Description: as for outcome 5
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL*hr
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 25
pg/mL*hr
  Cycle 2 (EE/norgestimate alone) | 16800 (5120)
  Cycle 3 (EE/norgestimate with erenumab): number analyzed (Participants) | 22
  Cycle 3 (EE/norgestimate with erenumab) | 16900 (4200)
Statistical Analysis 1: Comparison: Erenumab 140 mg + Estrogen/Progestin Contraceptive; [analysis description as in outcome 2, analysis 1]; Test type: Other; Least Squares Geometric Mean Ratio = 1.02, 90% CI 2-sided [0.94 to 1.12] — Ratio of EE/norgestimate + erenumab to EE/norgestimate alone

7. Secondary Outcome: Time to Reach the Maximum Concentration (Tmax) of Ethinyl Estradiol
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 25
hours
  Cycle 2 (EE/norgestimate alone) | 1.0 [1.0 to 2.0]
  Cycle 3 (EE/norgestimate with erenumab): number analyzed (Participants) | 22
  Cycle 3 (EE/norgestimate with erenumab) | 1.0 [1.0 to 1.8]

8. Secondary Outcome: Time to Reach the Maximum Concentration (Tmax) of Norgestrel
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 25
hours
  Cycle 2 (EE/norgestimate alone) | 1.5 [0.5 to 6.0]
  Cycle 3 (EE/norgestimate with erenumab): number analyzed (Participants) | 22
  Cycle 3 (EE/norgestimate with erenumab) | 1.5 [1.0 to 6.0]

9. Secondary Outcome: Time to Reach the Maximum Concentration (Tmax) of Norelgestromin
Description: as for outcome 5
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 25
hours
  Cycle 2 (EE/norgestimate alone) | 1.0 [0.5 to 4.0]
  Cycle 3 (EE/norgestimate with erenumab): number analyzed (Participants) | 22
  Cycle 3 (EE/norgestimate with erenumab) | 1.0 [0.5 to 4.0]

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: A treatment-related adverse event (AE) is any treatment-emergent AE that per investigator review has a reasonable possibility of being caused by the study drug.
  A device-related AE is any treatment-emergent AE that per investigator review has a reasonable possibility of being caused by the device (prefilled syringe) used to administer study drug.
Time Frame: From administration of erenumab on study day 66 through the end of the follow-up period on study day 150 (up to 84 days).
Population: The safety analysis set consisted of all participants who received at least one dose of study drug (erenumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 24
Participants
  All treatment-emergent adverse events | 17
  Serious adverse events | 0
  Fatal adverse events | 0
  Treatment-related adverse events | 2
  Treatment-related serious adverse events | 0
  Device-related adverse events | 1
  Device-related serious adverse events | 0

11. Secondary Outcome: Number of Participants Who Developed Anti-erenumab Binding Antibodies
Description: Blood samples were assessed for anti-erenumab binding antibodies. Samples testing positive for binding antibodies were also tested for neutralizing antibodies.
Time Frame: Baseline and day 150
Population: The safety analysis set consisted of all participants who received at least one dose of study drug (erenumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Number analyzed (Participants) | 24
Participants
  Binding antibody positive | 2
  Neutralizing antibody positive | 1

ADVERSE EVENTS:
Time Frame: From administration of erenumab on study day 66 through the end of the follow-up period on study day 150 (up to 84 days).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Erenumab 140 mg + Estrogen/Progestin Contraceptive
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 13/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab 140 mg + Estrogen/Progestin Contraceptive (N=24)
Nausea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 4
Headache (Nervous system disorders) | 8
Migraine (Nervous system disorders) | 2
Breast pain (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.